CLINICAL TRIAL: NCT04478110
Title: Community-Based Participatory Intervention to Improve Colorectal Cancer Screening Among Under-Served Korean Americans
Brief Title: Korean CRC Screening Study PT13599
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: Korean CRC; U54CA153513 (NIH)
Record Dates: First submitted 2020-07-15; First posted 2020-07-20 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Referral and Consultation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interactive education with linkage to care (Experimental): Main intervention components included interactive group education, navigation services and engagement of health care providers for referrals, and linkage to care
  Interventions: Behavioral: interactive group education, navigation services and engagement of health care providers for referrals, and linkage to care.
- general health education (Active Comparator): Receive a group education session focused on general health education and primary prevention issues.
  Interventions: Behavioral: Education Session on General Health

INTERVENTIONS:
Behavioral: interactive group education, navigation services and engagement of health care providers for referrals, and linkage to care. — The interactive group education was aimed to increase participant overall understanding of CRC, screening methods, and utilization of available resources such as home test kit and navigation services, with the ultimate goal of increasing screening rates. Clinical partners provided clinical support and ensured successful screening assessment and follow-ups by offering more flexible hours of clinic operation with bilingual medical staff on site. Patient navigation assistance was also offered based on participants' needs. The range of assistance included scheduling appointments with clinical partners for sigmoidoscopy/colonoscopy for screening and diagnosis after a FIT positive result, assisting paper.
  Arms: Interactive education with linkage to care
Behavioral: Education Session on General Health — Participants in the control group received a group education session in a similar format with that of the intervention group delivered by trained Korean community health educators. Different from the intervention group, the education focused on general health education and primary prevention issues, including routine health examinations and screening for various diseases such as cancer. Korean version of work and communication with a physician, and arranging transportation. standard printed materials and guidelines related to the education contents were also provided, including CRC screening guidelines.
  Arms: general health education

SUMMARY:
Korean Americans report the lowest and declined rates of colorectal cancer (CRC) screening, compared to general population in the United States. The present study aimed to evaluate the efficacy of a community-based multifaceted intervention designed to improve CRC screening among Korean Americans.

ELIGIBILITY:
Inclusion Criteria:

* Participants were eligible to participate in this study if they:

  1. were self-identified Korean Americans;
  2. were 50 years and older;
  3. did not have a colorectal polyp, CRC cancer, or a family history of CRC (first degree relative); and
  4. non-adherent to CRC screening guidelines (never had any CRC screening or were overdue for screening).

     Exclusion Criteria:

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 925 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
CRC screening rates | 12 months
  the completion of either FIT kit, sigmoidoscopy, or colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Grace X Ma, PhD, Principal Investigator — Temple University
Locations (1):
- Center for Asian Health, Lewis Katz School of Medicine, Temple University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Ma GX, Lee M, Beeber M, Das R, Feng Z, Wang MQ, Tan Y, Zhu L, Navder K, Shireman TI, Siu P, Rhee J, Nguyen MT. Community-Clinical Linkage Intervention to Improve Colorectal Cancer Screening Among Underserved Korean Americans. Cancer Health Disparities. 2019;3:e1-e15. Epub 2019 Aug 19. PMID 31528846
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC6746426/